CLINICAL TRIAL: NCT07358650
Title: A Multicenter, First-in-Human Clinical Study Evaluating the Safety and Performance of the MIST Device for Intraocular Pressure Reduction in Patients With Primary Open-Angle Glaucoma
Brief Title: Clinical Study Evaluating the Safety and Performance of the MIST Device for Intraocular Pressure Reduction in Patients With Primary Open-Angle Glaucoma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hexiris Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 020-3028
Record Dates: First submitted 2026-01-14; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Primary Open Angle Glaucoma
Keywords: scleral trephine; surgical trabeculectomy; bleb-forming intervention
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Intervention Model Description: Prospective, multicenter, open-label, non-randomized, single-arm, first-in-human clinical study: MIST + MMC: Subconjunctival MMC (0.02-0.04%) MMC will be injected subconjunctivally using a sterile technique, either prior to or following the procedure, at the surgeon's discretion.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- device intervention (Experimental): treatment with Hexiris MIST
  Interventions: Device: Hexiris Microinvasive Scleral Trephine (MIST)

INTERVENTIONS:
Device: Hexiris Microinvasive Scleral Trephine (MIST) — The punch needle of the Hexiris MIST device was designed to be injected securely into the conjunctiva/sclera and remove a core of tissue, creating a channel in the sclera of the eye for reduction of IOP.
  Other Names: subconjunctival mitomycin C injection

SUMMARY:
It is an interventional study for the treatment of Primary Open-Angle Glaucoma (POAG) using the Hexiris Microinvasive Scleral Trephine (MIST) system. This medical device includes a sclerectomy punch and injector assembly. It is a multicenter, open-label, non-randomized, single-arm study. Adults aged 40 years or more will be enrolled if the POAG is inadequately controlled by topical drug therapies. Only one eye per subject will be treated. The study will be performed on the first five patients in the operating room and the subsequent 20 patients will be treated under a slit-lamp in an aseptic environment (external patient clinic).Once treated with the MIST device, patients will return the next day, 1 week later and 1, 2, 3, 6, 9 and 12 months later. During these follow-up visits, the ophthalmologist will examine the eye and take measurements of the intraocular pressure.

DETAILED DESCRIPTION:
It is an interventional study for the treatment of Primary Open-Angle Glaucoma (POAG) using the Hexiris Microinvasive Scleral Trephine (MIST) system in adults aged 40 years or more. The primary goal of this new treatment is to reduce intraocular pressure in the affected eye.

The first five cases will be performed in the operating room. Safety data, including any serious adverse events occurring on Day 0 (surgery), will be reviewed by the safety monitor, who will issue a formal decision indicating whether the study may transition to the slit lamp or must continue in the operating room for the 20 subsequent patients.

The surgical technique is performed ab externo under topical anesthesia at the slit lamp.

Patients will be treated using the Hexiris MIST device along with a subconjunctival injection of mitomycin C (0.02-0.04%) using a sterile technique. There is postoperative care using topical antibiotics and steroids. The follow-up duration is 12-months post treatment with the Hexiris MIST device.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 40 years with uncontrolled mild to moderate POAG.
* IOP ≥ 18 mmHg on ≥1 topical IOP-lowering medications.
* Open angle on gonioscopy
* Clear cornea and healthy ocular surface
* Capable of giving informed consent, willingness to participate in the trial, and adhering to follow-up
* Glaucomatous visual field loss in one or both eyes at presentation on any of these criteria:

  * Reproducible and reliable visual field defects on 2 consecutive fields
  * Mild, moderate or advanced disease on mean deviation according to Hodapp classification
  * Healthy, mobile conjunctiva in the target quadrant (superior bulbar region)
  * Best-corrected Snellen visual acuity of 20/100 or better
  * Visual field mean deviation no worse than -18.0 dB (without dense paracentral scotomas)
* No anticipated need for other ocular surgeries (e.g., cataract) within 3 months of post-enrollment

Exclusion Criteria:

* Prior glaucoma filtering surgery (trabeculectomy, shunt or valve) in the treatment quadrant
* Angle-closure, neovascular, uveitic, or traumatic glaucoma.
* Eyes with conjunctival scarring, prior conjunctival surgery or other pathologies in the treatment quadrant
* Eyes with scleral thinning, staphyloma, or structural abnormalities in the treatment quadrant
* Uncontrolled IOP > 35 mmHg at screening.
* Active ocular infection or inflammation (e.g. blepharitis, conjunctivitis, keratitis, uveitis).
* Active or recent (within 6 months) iris neovascularization in the treatment quadrant
* Impaired episcleral venous drainage
* Anterior chamber intraocular lens
* Patients with uncontrolled bleeding disorders or those receiving anticoagulation therapy without appropriate perioperative management
* Advanced glaucomatous optic neuropathy.
* Fuchs endothelial dystrophy with clinical signs of endothelial decompensation.
* Central corneal thickness (CCT) > 600 μm.
* Pathological myopia.
* Patients unable to comply with postoperative follow-up or treatment instructions
* Women who are (i) pregnant, (ii) nursing, (iii) planning a pregnancy and (iv) of childbearing potential not using a reliable method of contraception as outlined below are excluded:

  * Hormonal methods and the intrauterine device (IUD) must be in use at least 30 days prior to first study drug administration
  * Barrier methods must be in use at least 14 days prior to study drug administration
  * Your male partner vasectomy must be completed 3 months prior to first study drug administration or a sperm count of 0 should be confirmed.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2026-01-15 (Actual); Primary Completion 2027-02-15 (Estimated); Study Completion 2027-03-15 (Estimated)

PRIMARY OUTCOMES:
Intraocular pressure lowering | change from baseline to Month 6
  Mean reduction in IOP (Goldmann applanation tonometry)

SECONDARY OUTCOMES:
Greater or equal to 20% reduction in intraocular pressure (IOP) | change from baseline to Months 6 and 12.
  Proportion of patients achieving ≥20% IOP reduction
Surgical success | at Month 12
  IOP 6-18 mmHg at Month 12 without additional surgery.
concomitant glaucoma medications | change from baseline at week 1 and Months 1, 2, 3, 6, 9 and 12.
  Change in the number of glaucoma medications
Composite surgical success | at Month 12
  IOP ≤ 21 mmHg and ≥20% reduction at Month 12 without additional glaucoma surgery, or clinically significant hypotony.
Bleb morphology | at week 1 and Months 1, 2, 3, 6, 9 and 12.
  Bleb morphology and stability - 4 point grading: healthy; injected; diffused bleb; others.
Corneal thickness | change from baseline to Month 6.
  Central corneal thickness (CCT) changes
Complications | at Day 1, week 1 and Months 1, 2, 3, 6, 9 and 12.
  Incidence of conjunctival erosion, hypotony-related complications (reported separately as numerical hypotony [IOP ≤ 5 mmHg] and clinical hypotony with complications).
Patients requiring Mitomycin C post treatment | at Day 1, week 1 and Months 1, 2, 3, 6, 9 and 12.
  Number of patients needing MMC injection after surgery.
Mitomycin C injection post treatment | at Day 1, week 1 and Months 1, 2, 3, 6, 9 and 12.
  Number of MMC injections needed post op per patient.
Safety - adverse events and device failures | day of surgery and at Day 1, week 1 and Months 1, 2, 3, 6, 9 and 12.
  reporting of adverse events and serious adverse events

CONTACTS AND LOCATIONS:
Locations (5):
- Canada (5):
  - Eye Care Centre NB, Dieppe, New Brunswick
  - Miramichi EyeNB & Surgical Centres of Excellence, Miramichi, New Brunswick
  - Prism Eye Institute Inc., Brampton, Ontario
  - Institut de l'oeil des Laurentides, Boisbriand, Quebec
  - Ophthalmology Clinic Bellevue, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No